CLINICAL TRIAL: NCT00111345
Title: Multicenter Therapy-Optimization Trial AML-BFM 2004 for the Treatment of Acute Myeloid Leukemias in Children and Adolescents
Brief Title: Therapy-Optimization Trial for the Treatment of Acute Myeloid Leukemias (AML) in Children and Adolescents
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BfArM 4022064; DKH 50-2728; NCT00478153 (obsolete NCT alias)
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-03

CONDITIONS: Myeloid Leukemia
Keywords: Acute; myeloid; leukemia; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia; Leukemia, Myeloid, Acute | interventions — Anthracyclines; Idarubicin; Daunorubicin; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Daunoxome, standard risk
  Interventions: Drug: liposomal daunorubicin
- 2 (Active Comparator): Idarubicin, standard risk
  Interventions: Drug: Anthracyclines
- 3 (Experimental): Daunoxome, high-risk, 2-CDA
  Interventions: Drug: 2-CDA
- 4 (Active Comparator): Idarubicin, high-risk, nothing
  Interventions: Drug: AI

INTERVENTIONS:
Drug: Anthracyclines — 3x12 mg/qm
  Other Names: Idarubicin
  Arms: 2
Drug: liposomal daunorubicin — 3x80 mg/qm
  Other Names: Daunoxome
  Arms: 1
Drug: 2-CDA — 2x6 mg/qm
  Other Names: Cladribine
  Arms: 3
Drug: AI — AI
  Arms: 4

SUMMARY:
Due to progressive therapy intensification in the four consecutive studies AML-BFM 78, 83, 93 and 98, prognosis for children with acute myeloid leukemia (AML) has improved steadily. In spite of the intensified therapy, rates of morbidity and mortality have remained unchanged or have even decreased. Against the background that about 40% of the patients still die from immediate causes of an underlying disease relapse or of nonresponse, it seems to be justifiable to intensify therapy - especially for high-risk patients - which on its parts will require an optimization of supportive measures. As the present risk stratification into standard- (SR) and high-risk (HR) patients has proved effective, we will pursue the risk-adapted therapy strategy.

The aim of the study is to improve prognosis in children with AML by intensification of cytostatic therapy and to evaluate by randomisation the equivalence of a prophylactic central nervous system (CNS) irradiation with a total dose of 18 Gy versus 12 Gy.

DETAILED DESCRIPTION:
During the last decade, prognosis in acute myelogenous leukemia (AML) in childhood has improved considerably, but still 30% of the children experience a relapse of disease and further 10% fail to respond sufficiently to the present therapies. A further intensification of therapy might improve the overall survival of these children, but possible, implicit side effects have to be considered carefully. Increase in dose intensification of the proven, effective anthracyclines will be limited by the risk of cumulative cardiotoxicity. A liposomal formulation of daunorubicin may offer a possibility to increase dosage, at least partially, without causing cumulative cardiotoxicity. Objective one of this randomised study is to ascertain if this dose increase improves therapy response and overall survival at acceptable toxicity. The previous experiences with liposomal daunorubicin, gathered from the relapse studies AML-BFM Rez 97 and International Therapy Study Relapsed AML 2001/012 as well as from the pilot study AML-BFM 2002P, have shown that the induction therapy is feasible in clinical centers with experience in AML therapy without leading to a marked increase of toxicity or prolongation of granulocytopenia.

First results of study AML-BFM 98 have shown that the patients of the standard risk (SR) group did not benefit from an additional, second induction (HAM). On this account we did not reintroduce this second induction course in the present study AML-BFM 2004. However, SR patients will take part in the randomisation of initial therapy with a general view to achieving higher effectiveness.

For patients of the high-risk group, the administration of 2-chloro-2-deoxyadenosine (2-CDA) will be integrated in the first phase of consolidation to achieve an even higher intensification. It could be shown that 2-CDA possesses good antileukemic activity in pediatric and adult AML. In a phase-II study it could also be demonstrated that 2-CDA has good effectiveness in combination with cytarabine. Results of phase-II studies conducted at St. Jude Children's Hospital, Memphis, showed that 2-CDA has good effectiveness especially in children with monoblastic leukemias (FAB M4/M5). Consequently, this intensification for high-risk patients, who present in more than half of the cases with monoblastic leukemias (FAB M4/5), may allow further improvement of therapy for this cohort. The pilot study AML-BFM 2002P confirmed that the study design was practicable without increasing significantly the risk of higher toxicity. However, median duration of aplasia was significantly prolonged in comparison to that of the AI (cytarabine, idarubicin)-block. Objective two of this study is to determine by randomisation if an improvement of efficiency is possible.

Study AML-BFM 98 has already focussed on the question of whether or not doses of CNS irradiation of 12 Gy and 18 Gy are equivalent with regard to their capacity of reducing the risk of relapse. As the results of study AML-BFM 87 confirmed the necessity of CNS irradiation, but did not reveal the necessary minimum dose, this randomisation has been implemented in order to prevent, as far as possible, late sequelae of CNS irradiation by reducing the radiation dose (= objective three).

As the number of patients of study AML-BFM 98 was not sufficient to resolve this question, this randomised analysis has been extended for a second period and will therefore be continued in the current study AML-BFM-2004.

Besides the intensification of cytostatic therapy, study AML-BFM 2004 seeks to optimise the quality of supportive therapy by implementing measures of quality assurance. This demands an up-to-date, complete documentation of each therapy phase. In studies AML-BFM 93 and 98, about 12% of deaths were due to primary complications such as leukostasis syndrome, haemorrhage or severe infections (4%), infections in aplasia before achieving remission (4%) or infections in remission (4%). Maybe the lives of even more children will be saved in the future by improved standards for the prevention of primary complications. Further, the efficacy of chemotherapy could be improved by less delays in therapy which are often due to infections or other complications.

ELIGIBILITY:
Inclusion Criteria:

* Age from >0 to </=18 years
* De novo AML, including children with Down syndrome, primary myelosarcomas or acute mixed lineage leukemia/biphenotypic leukemia (predominantly myeloid)
* Admission to one of the member hospitals in Germany participating in the study AML-BFM 2004

Exclusion Criteria:

* Children with pre-existing syndromes (except Down syndrome)
* AML as secondary malignancy
* Accompanying diseases which do not allow therapy according to the protocol
* Pre-treatment for more than 14 days with another intensive induction therapy

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 550 (Actual)
Dates: Start 2004-03; Primary Completion 2012-03 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Event-free and absolute survival from the date of diagnosis concerning objective 1 and from the date of randomisation concerning objective 2 | 5 years
Concerning objective 3: Disease-free survival from the date of randomisation | 5 years

SECONDARY OUTCOMES:
Cardiotoxicity | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Creutzig, Prof. Dr. med., Principal Investigator — Medical School Hannover; Dirk Reinhardt, Prof. Dr. med., Principal Investigator — Medical School Hanover
Locations (1):
- University Children's Hospital Muenster, Department of Paediatric Haematology and Oncology, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Steidel E, Orhan E, Rasche M, Pigazzi M, Tregnago C, Hoffmeister LM, Walter C, Dworzak M, Muhlegger N, von Neuhoff N, Locatelli F, Reinhardt D, Schneider M. Prognostic Value of Molecular Genetic Measurable Residual Disease (MRD) Monitoring in Pediatric Acute Myeloid Leukemia Expressing KMT2A::MLLT10. Eur J Haematol. 2025 Nov;115(5):493-504. doi: 10.1111/ejh.70019. Epub 2025 Aug 13. PMID 40803346
- [Derived] Tramsen L, Salzmann-Manrique E, Bochennek K, Klingebiel T, Reinhardt D, Creutzig U, Sung L, Lehrnbecher T. Lack of Effectiveness of Neutropenic Diet and Social Restrictions as Anti-Infective Measures in Children With Acute Myeloid Leukemia: An Analysis of the AML-BFM 2004 Trial. J Clin Oncol. 2016 Aug 10;34(23):2776-83. doi: 10.1200/JCO.2016.66.7881. Epub 2016 Jun 6. PMID 27269945
- [Derived] Hassler A, Bochennek K, Gilfert J, Perner C, Schoning S, Creutzig U, Reinhardt D, Lehrnbecher T. Infectious Complications in Children With Acute Myeloid Leukemia and Down Syndrome: Analysis of the Prospective Multicenter Trial AML-BFM 2004. Pediatr Blood Cancer. 2016 Jun;63(6):1070-4. doi: 10.1002/pbc.25917. Epub 2016 Jan 27. PMID 26814618
- [Derived] Creutzig U, Zimmermann M, Bourquin JP, Dworzak MN, Fleischhack G, Graf N, Klingebiel T, Kremens B, Lehrnbecher T, von Neuhoff C, Ritter J, Sander A, Schrauder A, von Stackelberg A, Stary J, Reinhardt D. Randomized trial comparing liposomal daunorubicin with idarubicin as induction for pediatric acute myeloid leukemia: results from Study AML-BFM 2004. Blood. 2013 Jul 4;122(1):37-43. doi: 10.1182/blood-2013-02-484097. Epub 2013 May 23. PMID 23704089
- [Derived] Creutzig U, Zimmermann M, Bourquin JP, Dworzak MN, Fleischhack G, von Neuhoff C, Sander A, Schrauder A, von Stackelberg A, Ritter J, Stary J, Reinhardt D. CNS irradiation in pediatric acute myleoid leukemia: equal results by 12 or 18 Gy in studies AML-BFM98 and 2004. Pediatr Blood Cancer. 2011 Dec 1;57(6):986-92. doi: 10.1002/pbc.22955. Epub 2011 Apr 7. PMID 21480469
- [Derived] Klusmann JH, Creutzig U, Zimmermann M, Dworzak M, Jorch N, Langebrake C, Pekrun A, Macakova-Reinhardt K, Reinhardt D. Treatment and prognostic impact of transient leukemia in neonates with Down syndrome. Blood. 2008 Mar 15;111(6):2991-8. doi: 10.1182/blood-2007-10-118810. Epub 2008 Jan 8. PMID 18182574
- [Derived] Meyer LH, Queudeville M, Eckhoff SM, Creutzig U, Reinhardt D, Karawajew L, Ludwig WD, Stahnke K, Debatin KM. Intact apoptosis signaling in myeloid leukemia cells determines treatment outcome in childhood AML. Blood. 2008 Mar 1;111(5):2899-903. doi: 10.1182/blood-2007-08-109058. Epub 2007 Dec 14. PMID 18083847
- See also: Click here for more information about this study: Multicenter Therapy-Optimization Trial AML-BFM 2004 for the Treatment of Acute Myeloid Leukemias in Children and Adolescents — http://aml.mh-hannover.de/